CLINICAL TRIAL: NCT01687478
Title: A Study to Assess the Short-Term Efficacy and Safety of Olanzapine and Fluoxetine Compared to Placebo and Fluoxetine for Nonpsychotic Treatment-Resistant Depression
Brief Title: A Study of Olanzapine and Fluoxetine for Treatment-resistant Depression
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Interim assessment: Lack of efficacy
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13702; F1D-CR-HGNB (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-09-07; First posted 2012-09-19 (Estimated); Results first posted 2017-08-24 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-09

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Olanzapine; Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Olanzapine + Fluoxetine (Experimental): Olanzapine starting dose is 5 milligram (mg) (1 tablet). May titrate up to 10 mg (2 tablets), or 15 mg (3 tablets) administered once daily by mouth for 8 weeks.
  Fluoxetine starting dose is 20 mg. May titrate up to 40 mg or 50 mg administered once daily by mouth for 8 weeks.
  Interventions: Drug: Olanzapine; Drug: Fluoxetine
- Placebo + Fluoxetine (Placebo Comparator): Placebo matches the Olanzapine tablet for blinding.
  Fluoxetine starting dose is 20 mg, then may titrate up to 40 mg or 50 mg administered once daily by mouth for 8 weeks.
  Interventions: Drug: Fluoxetine; Drug: Placebo

INTERVENTIONS:
Drug: Olanzapine — Administered Orally
  Other Names: LY170053; Zyprexa
  Arms: Olanzapine + Fluoxetine
Drug: Fluoxetine — Administered Orally
  Other Names: LY110140; Prozac
Drug: Placebo — Administered Orally
  Arms: Placebo + Fluoxetine

SUMMARY:
The purpose of this study is to assess the efficacy and safety of olanzapine and fluoxetine compared to placebo and fluoxetine as treatment for treatment-resistant depression (TRD) in Chinese participants.

ELIGIBILITY:
Inclusion Criteria:

* Have single or recurrent unipolar major depressive disorder (MDD) without psychotic features by Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition-Text Revision (DSM-IV-TR) clinical assessment
* Have a total score ≥22 on the 17-item Hamilton Depression Rating Scale (HAM-D17) at screening and randomization
* Have treatment-resistant depression (TRD), defined as having failed to achieve a satisfactory antidepressant response, in the opinion of the investigator, to separate treatment courses of at least 2 different antidepressants, other than fluoxetine, of adequate dosage and duration (≥6 weeks) within the current major depressive episode

Exclusion Criteria:

* Have a diagnosis of Parkinson's disease or a related disorder
* Have a current or lifetime diagnosis of any of the following conditions, according to DSM-IV-TR criteria: Schizophrenia; Schizophreniform Disorder; Schizoaffective Disorder; Delusional Disorder; Psychotic Disorder Not Otherwise Specified; Bipolar Disorder I or II; Delirium of any type; Dementia of any type; Amnestic Disorder; any Substance-Induced Disorder; or any Psychotic Disorder due to a General Medical Condition
* Have a current diagnosis of post-partum depression or MDD with a seasonal pattern as defined in the DSM-IV-TR
* Have paranoid, schizoid, schizotypal, antisocial, or borderline personality disorder (Axis II) as a comorbid or primary diagnosis, based on DSM-IV-TR criteria
* Have DSM-IV-TR substance dependence/abuse or are not willing to avoid use of the substance (not including dependence on nicotine or caffeine) within 30 days of screening
* Are actively suicidal in the judgment of the investigator
* Have uncorrected narrow-angle glaucoma
* Have had one or more seizures without a clear and resolved etiology
* Have leukopenia
* Have any acute, serious, or unstable medical conditions
* Have an increased serum prolactin concentration at screening
* Have a rate-corrected cardiac QT interval, calculated using Bazett's formula (QTc Bazett's [Rate-corrected cardiac QT interval on electrocardiogram calculated using Bazett's formula(QTcB)]), on Electrocardiogram (ECG) >450 milliseconds (male) or >470 milliseconds (female) at screening
* Have a history of allergic reaction to olanzapine, fluoxetine, or olanzapine in combination with fluoxetine
* Have had treatment with olanzapine, fluoxetine, or olanzapine in combination with fluoxetine withdrawn due to clinically significant and/or intolerable adverse effects within 6 months of screening
* Have received treatment with remoxipride within 6 months of randomization
* Have received treatment with depot antipsychotics within one dosing interval before randomization
* Have received electroconvulsive therapy (ECT) or vagus nerve stimulation (VNS) treatment within the current MDD episode, or has a history of failure to respond to adequate treatment courses of ECT or VNS, or is expected to require ECT or VNS at any time during the study
* Have received previous treatment with clozapine
* Have received treatment with a monoamine oxidase inhibitor (MAOI) within 14 days of screening, or are expected to need MAOI treatment at any time during the study or up until 5 weeks after study discontinuation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2012-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (11):
- China (11):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baoding
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beijing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Changsha
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guangzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hangzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kunming
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nanjing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shanghai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wuhan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Xi'an
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Xinxiang

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Olanzapine + Fluoxetine: Olanzapine starting dose is 5 milligram (mg). May titrate up to 10 mg, or 15 mg administered once daily by mouth for 8 weeks.
  Fluoxetine starting dose is 20 mg. May titrate up to 40 mg or 50 mg administered once daily by mouth for 8 weeks.
Period: Overall Study
Arm/Group | Olanzapine + Fluoxetine | Placebo + Fluoxetine
Started | 88 | 88
Safety Analysis Set | 88 | 87
Completed | 56 | 49
Not Completed | 32 | 39
Not completed — Adverse Event | 3 | 10
Not completed — Lost to Follow-up | 1 | 3
Not completed — Protocol Violation | 0 | 2
Not completed — Withdrawal by Subject | 21 | 19
Not completed — Physician Decision | 1 | 3
Not completed — Entry Criteria Not Met | 6 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Olanzapine + Fluoxetine | Placebo + Fluoxetine | Total
Number analyzed (Participants) | 88 | 88 | 176
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.63 (12.18) | 41.45 (12.44) | 40.04 (12.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 36 | 77
  Male | 47 | 52 | 99
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 88 | 88 | 176
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 88 | 88 | 176
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 88 | 88 | 176
Montgomery-Äsberg Depression Rating Scale (MADRS) Total Score [Mean (Standard Deviation); unit: units on a scale] — The MADRS is a rating scale for severity of depressive mood symptoms. The MADRS has a 10-item checklist. Items are rated on a scale of 0-6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms).
  units on a scale | 32.1 (5.3) | 31.8 (4.8) | 32.0 (5.0)
17 Item Hamilton Rating Scale for Depression (HAM-D17) Total Score [Mean (Standard Deviation); unit: units on a scale] — The 17-item HAMD measures depression severity. Each item was evaluated and scored using either a 5-point scale (e.g. absent, mild, moderate, severe, very severe) or a 3-point scale (e.g. absent, mild, marked). The total score of HAMD-17 may range from 0 (normal) to 52 (severe).
  units on a scale | 24.6 (2.6) | 25.0 (2.6) | 24.8 (2.6)
Clinical Global Impressions-Severity of Depression (CGI-S) [Mean (Standard Deviation); unit: units on a scale] — The CGI-S measures severity of illness at the time of assessment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill participants).
  units on a scale | 4.9 (0.6) | 4.9 (0.7) | 4.9 (0.7)
Age of First Major Depressive Disorder (MDD) Episode [Mean (Standard Deviation); unit: years] | 29.92 (12.61) | 34.07 (12.69) | 30.00 (12.79)
Years Since the First MDD Episode [Mean (Standard Deviation); unit: years] | 8.71 (6.21) | 7.38 (7.86) | 8.05 (7.10)
Years Since the Most Recent MDD Episode [Mean (Standard Deviation); unit: years] | 3.66 (5.12) | 3.23 (4.15) | 3.45 (4.65)
Number of Previous Lifetime MDD Episodes [Mean (Standard Deviation); unit: Number of MDD Episodes] | 1.4 (1.4) | 1.3 (2.1) | 1.3 (1.8)
Number of Previous MDD Episodes Within the Last 36 Months [Mean (Standard Deviation); unit: Number of MDD Episodes] | 0.5 (0.8) | 0.5 (1.1) | 0.5 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to 8 Week Endpoint in Montgomery-Äsberg Depression Rating Scale (MADRS)
Description: The MADRS total score is the sum of the 10 items; therefore the possible MADRS total score ranges from 0 to 60. A higher MADRS total score indicates a greater severity of depressive symptoms. Least square means (LSM) change from baseline, standard error was derived using mixed model repeated measures (MMRM) methodology with factors for treatment, Pooled Investigator, Visit, (Baseline + Treatment)*Visit.
Time Frame: Baseline, 8 Weeks
Population: Participants in the full analysis set (FAS) population: all randomized participants who had a baseline and at least one post-baseline MADRS total score measurement.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Olanzapine + Fluoxetine | Placebo + Fluoxetine
Number analyzed (Participants) | 87 | 86
Units on a scale | -15.92 (1.20) | -14.30 (1.28)
Statistical Analysis 1: Comparison: Olanzapine + Fluoxetine vs Placebo + Fluoxetine; Test type: Superiority or Other; Mean Difference (Net) = -1.62, 95% CI 2-sided [-5.04 to 1.80] — The Confidence Interval is based on the treatment difference LS Mean changes from baseline between Olanzapine + Fluoxetine and Placebo + Fluoxetine

2. Secondary Outcome: Mean Change From Baseline to 8 Week Endpoint in Clinical Global Impressions-Severity of Depression (CGI-S) Scale
Description: CGI-S scale measures severity of illness at the time of assessment compared with start of treatment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill participants). The LS mean (LSM) change from baseline, standard error was derived using MMRM methodology with factors for treatment , Pooled Investigator , Visit , (Baseline + Treatment)*Visit.
Time Frame: Baseline, 8 Weeks
Population: Participants in the FAS population: all randomized participants who had a baseline and at least one post-baseline MADRS total score measurement.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Olanzapine + Fluoxetine | Placebo + Fluoxetine
Number analyzed (Participants) | 87 | 86
Units on a scale | -1.43 (0.15) | -1.63 (0.16)

3. Secondary Outcome: Mean Change From Baseline to 8 Week Endpoint in the Simpson-Angus Scale (SAS)
Description: SAS scale consists of 10 items including 7 items that address bradykinesia-rigidity and additional single items for tremor, glabellar tap,and salivation. Each item represents a specific physical condition and is rated on a 5-point category rating scale ranging from 0 (complete absence of the condition) to 4 (the condition is present to an extreme degree).The total score is obtained by adding the scores for the 10 individual items making the maximum possible score is 40. Higher scores are indicative of more severe Parkinsonian-type symptoms.
Time Frame: Baseline, 8 Weeks
Population: All randomized participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Olanzapine + Fluoxetine | Placebo + Fluoxetine
Number analyzed (Participants) | 88 | 87
units on a scale | 0.03 (1.71) | -0.14 (1.72)

4. Secondary Outcome: Mean Change From Baseline to 8 Week Endpoint in the Short-Form 36 Health Survey (SF-36)
Description: SF-36, version 2 is a generic participant-rated questionnaire and consists of 36 questions covering the following 8 health domains (subscales): general health, role limitations because of physical problems, role limitations due to emotional problems, physical functioning, bodily pain, mental health, social functioning, and vitality. Each subscale is scored by summing the individual items and transforming the scores into a 0 to 100 scale, with higher scores indicating better health status or functioning. Two summary scores, the physical component summary (PCS) and the mental component summary (MCS) were constructed based on the eight SF-36 subscales. Both PCS and MCS range from 0-100 with higher scores indicating better health or functioning.
Time Frame: Baseline, 8 Weeks
Population: All randomized participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Olanzapine + Fluoxetine | Placebo + Fluoxetine
Number analyzed (Participants) | 88 | 88
units on a scale
  Physical Functioning | 2.20 (7.51) | 0.70 (7.47)
  Role-Physical | 3.99 (11.79) | 3.93 (11.23)
  Bodily Pain | 6.81 (12.05) | 0.02 (11.30)
  General Health | 5.82 (11.49) | 2.84 (9.44)
  Vitality | 7.43 (13.54) | 5.04 (9.83)
  Social Functioning | 6.13 (13.55) | 4.56 (11.78)
  Role-Emotional | 6.61 (12.39) | 6.71 (12.12)
  Mental Health | 8.98 (13.46) | 8.43 (11.99)
  Mental Component Score | 8.87 (14.29) | 8.73 (12.54)
  Physical Component Score | 2.87 (7.59) | -0.65 (7.22)

5. Secondary Outcome: Mean Change From Baseline to 8 Week Endpoint in the Sheehan Disability Scale (SDS)
Description: SDS consists of 3 items (work/school, social life/leisure activities, and family life/home responsibilities). Total scores range from 0 to 30 with higher values indicating greater disruption. Individual Item scores range from 0 to 10 with higher values indicating greater disruption.
Time Frame: Baseline, 8 Weeks
Population: All randomized participants.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Olanzapine + Fluoxetine | Placebo + Fluoxetine
Number analyzed (Participants) | 88 | 88
Units on a scale
  Work/School (n=68,65) | -1.34 (2.71) | -1.55 (2.89)
  Social Life (n=79,79) | -1.70 (2.66) | -1.49 (2.85)
  Family Life (n=79,78) | -1.63 (3.00) | -1.53 (2.66)
  SDS Total Score (68,64) | -4.57 (7.75) | -4.41 (7.89)

6. Secondary Outcome: Percentage of Participants Who Achieve a Response Based on a ≥50% Reduction From Baseline in MADRS Total Score
Description: The MADRS total score is the sum of the 10 items; therefore the possible MADRS total score ranges from 0 to 60. A higher MADRS total score indicates a greater severity of depressive symptoms.
Time Frame: Baseline,8 Weeks
Population: All randomized participants who had a baseline and at least one post-baseline MADRS total score measurement.
Measure: Number; unit: Percent of participants
Arm/Group | Olanzapine + Fluoxetine | Placebo + Fluoxetine
Number analyzed (Participants) | 87 | 86
Percent of participants | 65.5 | 61.2

7. Secondary Outcome: Percentage of Participants Who Achieve Remission Based on MADRS Total Score ≤10 at 8 Weeks
Description: The MADRS consists of 10 items with each item rated on a scale ranging from 0 to 6. Fixed descriptors appear along the scale for each item at points 0, 2, 4, and 6, to standardize the gradation of response along the scale. The MADRS total score is the sum of the 10 items; therefore the possible MADRS total score ranges from 0 to 60. A higher MADRS total score indicates a greater severity of depressive symptoms.
Time Frame: Baseline, 8 Weeks
Population: All randomized participants who had a baseline and at least one post-baseline MADRS total score measurement.
Measure: Number; unit: Percent of participants
Arm/Group | Olanzapine + Fluoxetine | Placebo + Fluoxetine
Number analyzed (Participants) | 87 | 86
Percent of participants | 37.9 | 38.8

8. Secondary Outcome: Mean Change From Baseline to 8 Week Endpoint in the Barnes Akathisia Scale (BAS)
Description: BAS is used to rate observable, restless movements of drug induced akathisia and the subjective awareness of restlessness and any distress associated with the akathisia. The BAS consists of the following 3 items: an objective assessment of akathisia symptoms; a subjective assessment of the patient's awareness of inner restlessness; and a global clinical assessment of akathisia. The first two items are rated on a 4-point scale ranging from 0 (no abnormal movements or the absence of inner restlessness) to 3 (severe akathisia or the awareness of intense compulsion to move most of the time). The last item, the global clinical assessment of akathisia, is rated on a 5-point scale, ranging from 0 (no evidence of akathisia) to 5 (severe akathisia). Total BAS score ranges from 0 to 14 with a higher score representing worse results.
Time Frame: Baseline, 8 Weeks
Population: All randomized participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Olanzapine + Fluoxetine | Placebo + Fluoxetine
Number analyzed (Participants) | 88 | 87
units on a scale | -0.01 (2.24) | -0.04 (2.13)

9. Secondary Outcome: Mean Change From Baseline to 8 Week Endpoint in the Abnormal Involuntary Movement Scale (AIMS)
Description: AIMS is a 12-item scale. Items 1 to 8 are rated on a 5-point scale ranging from 0 (no dyskinetic movements) to 4 (severe dyskinetic movements). Item 9 assesses the participant's incapacitation due to abnormal movements, and item 10 assesses the participant's awareness of the abnormal movements and associated distress. Items 9 and 10 are rated on 5-point scales ranging from 0 (none or no awareness) to 4 (severe or aware, severe distress). Items 11 and 12 are yes/no questions regarding the dental status of the participant. The total score is the sum of the scores for the 12 items and the possible total score ranges from 0 to 42. A higher total score is indicative of more severe dyskinetic movements.
Time Frame: Baseline, 8 Weeks
Population: All randomized participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Olanzapine + Fluoxetine | Placebo + Fluoxetine
Number analyzed (Participants) | 88 | 87
units on a scale | -0.16 (1.47) | -0.31 (3.28)

ADVERSE EVENTS:
Description: All participants in the safety analysis set.
Arm/Group | Olanzapine + Fluoxetine | Placebo + Fluoxetine
Serious Adverse Events (participants affected / at risk) | 1/88 | 1/87
Other Adverse Events (participants affected / at risk) | 55/88 | 45/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olanzapine + Fluoxetine (N=88) | Placebo + Fluoxetine (N=87)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Olanzapine + Fluoxetine (N=88) | Placebo + Fluoxetine (N=87)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Cardiovascular insufficiency (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 2 (2) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 4 (4)
Retching (Gastrointestinal disorders) | 0 (0) | 1 (1)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tongue disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 2 (2) | 3 (3)
Chest discomfort (General disorders) | 1 (1) | 2 (2)
Chest pain (General disorders) | 1 (1) | 0 (0)
Discomfort (General disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 3 (3) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Hunger (General disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0)
Sensation of foreign body (General disorders) | 0 (0) | 1 (1)
Thirst (General disorders) | 2 (2) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 6 (6) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 7 (7) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 5 (5) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 2 (2)
Blood cholesterol increased (Investigations) | 5 (5) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 1 (1)
Blood glucose increased (Investigations) | 2 (2) | 1 (1)
Blood pressure increased (Investigations) | 2 (2) | 0 (0)
Blood prolactin increased (Investigations) | 9 (9) | 2 (2)
Blood triglycerides increased (Investigations) | 7 (7) | 3 (3)
Electrocardiogram abnormal (Investigations) | 1 (1) | 1 (1)
Electrocardiogram t wave abnormal (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 3 (3) | 0 (0)
High density lipoprotein decreased (Investigations) | 1 (1) | 1 (1)
Lipids increased (Investigations) | 3 (3) | 0 (0)
Low density lipoprotein increased (Investigations) | 3 (3) | 1 (1)
Transaminases increased (Investigations) | 3 (3) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 4 (4)
Weight increased (Investigations) | 8 (8) | 2 (2)
White blood cell count decreased (Investigations) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 6 (6) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/41 (0) | 1/35 (1)
Akathisia (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 5 (5)
Extrapyramidal disorder (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 3 (3)
Hypokinesia (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 15 (17) | 3 (4)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (2) | 0 (0)
Dysphoria (Psychiatric disorders) | 0 (0) | 1 (1)
Fear (Psychiatric disorders) | 1 (1) | 0 (0)
Initial insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Mental disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Nervousness (Psychiatric disorders) | 2 (2) | 2 (3)
Restlessness (Psychiatric disorders) | 2 (2) | 3 (3)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Somatic delusion (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 1 (1)
Urine odour abnormal (Renal and urinary disorders) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days